CLINICAL TRIAL: NCT00997841
Title: Conventional Versus Point-of-care Based Coagulation Management in Cardiac Surgery Patients Suffering From Increased Bleeding Tendency - a Prospective and Randomized Study
Brief Title: Conventional Versus Point-of-care Based Coagulation Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Dr. Christian Weber, Goethe University Frankfurt, Clinic for Anaesthesiology, Theodor Stern Kai 7, 60590 Frankfurt am Main, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: POC-9509
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2009-10

CONDITIONS: Cardiac Surgery; Coagulation Management
Keywords: POC; ROTEM; Multiplate; bleeding tendency; coagulation management; amount of transfused red blood cell concentrates,; FFP; platelet concentrates; rate of rethoracotomy; ventilation time
MeSH Terms: conditions — Hemostatic Disorders | interventions — Point-of-Care Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- POC algorithm (Active Comparator): cardiac surgery patients suffering from increased perioperative bleeding and being treated following Point of Care based algorithm
  Interventions: Procedure: Point-of-Care versus conventional coagulation management
- conventional algorithm (Active Comparator): cardiac surgery patients suffering from increased perioperative bleeding and being treated following conventional coagulation management algorithm
  Interventions: Procedure: Point-of-Care versus conventional coagulation management

INTERVENTIONS:
Procedure: Point-of-Care versus conventional coagulation management — Patients are randomized to receive either point-of-care based or conventional coagulation measurements based coagulation therapy in the case of increased perioperative bleeding tendency
  Other Names: ROTEM; Multiplate; Point-of-Care

SUMMARY:
The purpose of the study is to determine the efficacy of two different algorithms for coagulation management in patients undergoing cardiac surgery suffering from increased bleeding tendency. Algorithm 1 is based on conventional coagulation analyses (INR, aPTT, platelet count, fibrinogen concentration,...) and Algorithm 2 is based on thrombelastometry using the ROTEM-device and impedance aggregometry using the Multiplate device.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years, combined surgical procedures (ACB & valve surgery), double valve surgery, aortic surgery, Re-Dos

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
amount of transfused red blood cell concentrates | 24 h after begin of surgical intervention

SECONDARY OUTCOMES:
other transfused blood products including FFP, platelet concentrates and coagulation factor concentrates | 24h after surgical intervention
rate of rethoracotomy for bleeding | 24h after surgical intervention
ventilation time on ICU | till discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Weber, Dr., Principal Investigator — Johann Wolfgang Goethe University Frankfurt, Clinic for Anaesthesiology, Intensive Care Medicine and Pain Therapy
Locations (2):
- Germany (2):
  - University Hospital Essen, Clinic for Anesthesiology and Intensive Care Medicine, Essen
  - Johann Wolfgang Goethe University Frankfurt, Clinic for Anaesthesiology, Frankfurt am Main

REFERENCES:
- [Background] Görlinger K, Jambor C, Hanke A, Adamzik M, Hartmann M, Rahe-Meyer N. Thrombelastometry and impedance aggregometry based algorithm for coagulation management in cardiac surgery. Intensive Care Med 33: 196, 2007.
- [Background] Görlinger K, Jambor C, Hanke A, Adamzik M, Hartmann M, Rahe-Meyer N. Perioperative coagulation management and controll of platelet transfusion by point-of-care platelet function analysis. Transfus Med Hemother 34: 396-411, 2007.
- [Background] Görlinger K, Bergmann L, Hartmann M, Marggraf G, Kamler M, Müller-Beißenhirtz H. Reduction of blood transfusion rate by thrombelastometry and impedance aggregometry based point-of-care coagulation management in thoracic and cardiovascular surgery. Appl Cardiopulmon Pathophysiol 13: 174-7, 2009.
- [Derived] Weber CF, Gorlinger K, Meininger D, Herrmann E, Bingold T, Moritz A, Cohn LH, Zacharowski K. Point-of-care testing: a prospective, randomized clinical trial of efficacy in coagulopathic cardiac surgery patients. Anesthesiology. 2012 Sep;117(3):531-47. doi: 10.1097/ALN.0b013e318264c644. PMID 22914710